CLINICAL TRIAL: NCT03031509
Title: Treatment of Nonunion of Limb Fracture With Human Amniotic Epithelial Cells（hAECs）
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai East Hospital (Other)
Collaborators: Shanghai iCELL Biotechnology Co., Ltd, Shanghai, China (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DFSC-2017（CR）-01
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Nonunion Fracture
Keywords: Nonunion Fracture of limb
MeSH Terms: conditions — Fractures, Ununited | interventions — Debridement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hAECs treatment (Experimental): Human Amniotic Epithelial Cells of 50 million transplant to nonunion site after debridement surgery
  Interventions: Biological: Human Amniotic Epithelial Cells; Procedure: debridement
- debridement surgery (Sham Comparator): debridement surgery
  Interventions: Procedure: debridement

INTERVENTIONS:
Biological: Human Amniotic Epithelial Cells — Human Amniotic Epithelial Cells transplant after debridement
  Arms: hAECs treatment
Procedure: debridement — debridement

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of human amniotic epithelial cells transplant in nonunion of limb fracture patients.

DETAILED DESCRIPTION:
In this study, patients of nonunion after limb fracture will be treated with human amniotic epithelial cells. Clinical and radiological assessment is performed.

hAECs developing from the epiblast as early as 8 days after fertilization, recent data reported indicate that hAECs possess proper osteogenic differentiation potential and a localized modulatory influence on the early tissue remodeling process, making these cells a promising stem cell source for bone regeneration after fractures.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with nonunion of limbs by x-ray and bone scan;
* compliance to treatment and long term follow-up;
* be able and willing to participate in the study;
* written informed consent before study.

Exclusion Criteria:

* pregnant or breastfeeding;
* patients with malignancy, immunocompromised ( HIV AIDS, Diabetes mellitus, active Hepatitis), in a immunosuppressant therapy ( chemotherapy or steroids), OR health status, mental diseases, which will influence the study;
* patients undergoing any other treatment that are not related to this study;
* others considered not appropriate selected patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2018-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
time for bone union | 6 months
  Bone union was evaluated at 6-month after surgery according to the following definition.Definition of bone union is when simple X-ray findings reveal that bone trabeculae or cortical bone exceeds the fracture site.

SECONDARY OUTCOMES:
pain in fracture site | 1 year
limb functional score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: XIA LI, Dr., Principal Investigator — Shanghai East Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miki T, Lehmann T, Cai H, Stolz DB, Strom SC. Stem cell characteristics of amniotic epithelial cells. Stem Cells. 2005 Nov-Dec;23(10):1549-59. doi: 10.1634/stemcells.2004-0357. Epub 2005 Aug 4. PMID 16081662
- [Background] Si J, Dai J, Zhang J, Liu S, Gu J, Shi J, Shen SG, Guo L. Comparative investigation of human amniotic epithelial cells and mesenchymal stem cells for application in bone tissue engineering. Stem Cells Int. 2015;2015:565732. doi: 10.1155/2015/565732. Epub 2015 Mar 5. PMID 25834575
- [Background] Jiawen S, Jianjun Z, Jiewen D, Dedong Y, Hongbo Y, Jun S, Xudong W, Shen SG, Lihe G. Osteogenic differentiation of human amniotic epithelial cells and its application in alveolar defect restoration. Stem Cells Transl Med. 2014 Dec;3(12):1504-13. doi: 10.5966/sctm.2014-0118. Epub 2014 Nov 3. PMID 25368378